CLINICAL TRIAL: NCT06532201
Title: Effects of Su Jok Therapy on Pain, Fatigue, Nausea-Vomiting and Spiritual Well-Being Levels in Patients Receiving Chemotherapy
Brief Title: Effects of Su Jok Therapy on Pain, Fatigue, Nausea-Vomiting and Spiritual Well-Being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Güzel Nur Yıldız, Dr, Dr., Muş Alparslan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mus Alparslan U
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Chemotherapy
Keywords: su-jok; cancer patients; Pain; fatigue; nausea-vomiting; spiritual well-being
MeSH Terms: conditions — Neoplasms; Pain; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Su-jok Therapy Group /EXPERIMENTAL GROUP (Experimental): Su Jok will be applied to the reflection points on the hand based on the painful area of the individual. The painful areas will be determined with the applicator and black pepper seeds will be placed on these areas. Circular massage will be applied to the areas where the seeds are located for 30 minutes.
  Interventions: Other: Su jok seed therapy
- Control Group (No Intervention)

INTERVENTIONS:
Other: Su jok seed therapy — Su Jok will be applied to the reflection points on the hand based on the painful area of the individual. The painful areas will be determined with the applicator and black pepper seeds will be placed on these areas. Circular massage will be applied to the areas where the seeds are located for 30 minutes.
  Arms: Su-jok Therapy Group /EXPERIMENTAL GROUP

SUMMARY:
This study aims to examine the effects of sujok therapy on pain, fatigue, nausea-vomiting and spiritual well-being levels in patients receiving chemotherapy. The following questions are being answered;

* Does sujok therapy affect pain levels in cancer patients?
* Does sujok therapy affect fatigue levels in cancer patients?
* Does sujok therapy affect nausea-vomiting levels in cancer patients?
* Does sujok therapy affect spiritual well-being levels in cancer patients?

DETAILED DESCRIPTION:
Location of the study:

Research data will be collected in the oncology unit of Muş State Hospital.

Research universe, sample, research group:

The research universe will consist of patients who apply to the oncology service in the hospital where the study is conducted and receive treatment. It was determined that the required sample size for the study to exceed 80% with a 95% confidence interval, 0.05 significance level and medium effect size was 68 people, with 34 people in each group.

Data collection tools:

"Descriptive Characteristics Form" and "Visual Analog Scale-VAS", "Cancer Fatigue Scale", "Rhodes Nausea-Vomiting and Retching Index" and "Spiritual Well-Being Scale" will be used as data collection tools.

Descriptive Characteristics Form This form includes questions such as patients' age, gender, socioeconomic level, and educational status.

Visual Analog Scale-VAS: The severity of the symptom experienced by the patient is measured by marking a numbered point on this line. VAS markings are repeated before and during the procedure, regardless of the previous marking location. In this study, a 0-10 point scale will be used to evaluate the pain levels of individuals with VAS.

Cancer Fatigue Scale (KPSS): Its validity and reliability in Turkey was conducted by Şahin et al. in 2018. The scale, consisting of a total of 15 items and three sub-dimensions, has a 5-point Likert structure. The highest score that can be obtained from the scale is 60 points. It is stated that the higher the score, the higher the fatigue level. The internal consistency coefficient of the scale is 0.74.

Rhodes nausea-vomiting and retching index (NBSI): Its validity and reliability in Turkish was conducted by Tan and Genç. The scale, which has a five-point Likert structure (0= least distress level, 4= most distress), has eight items that measure the number and severity of nausea-vomiting-retching in the last 24 hours. The highest score that can be obtained from the scale is 32, and it is stated that the distress level increases as the score increases. The internal consistency coefficient of the scale is 0.95. Spiritual Well-Being Scale: Its Turkish adaptation was made by Aktürk et al. (2017). The scale was created to determine the spiritual well-being of cancer patients or individuals with other chronic diseases. The scale is a five-point Likert type and consists of 12 items. The items of the scale have a numbering system between 0 and 4 (0-Not at all, 4-A lot). The total score of the scale is 0-48 points. A higher scale score indicates better spiritual well-being. The total Cronbach alpha value of the scale is 0.87.

RANDOMIZATION Patients who apply to the oncology unit for chemotherapy will be numbered according to the order of application. Patients will be divided into experimental and control groups using the "RANDOMIZER" program.

Control group: No intervention will be made to this group. When participating in the study, participants will be asked to fill out the "Visual Analog Scale-VAS", "Cancer Fatigue Scale", "Rhodes Nausea-Vomiting and Retching Index" and "Spiritual Well-Being Scale" after one and two months.

Experimental group: Su jok therapy will be applied to this group using black pepper seeds. A total of 8 sessions (twice a week for 4 weeks) of therapy will be applied. Black pepper seeds will be placed on a certain point of the patient's hand and taped. After two hours, they will be asked to remove and throw away. When participating in the study, after one and two months, participants will be asked to fill out the "Visual Analog Scale-VAS", "Cancer Fatigue Scale", "Rhodes Nausea-Vomiting and Retching Index" and "Spiritual Well-Being Scale".

In the last stage, the data obtained will be compared within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being diagnosed with cancer
* Being receiving chemotherapy
* No communication problems

Exclusion Criteria:

* Deterioration or death during the research process
* Requesting to withdraw from the research
* Incomplete filling of forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
"VAS" will be used to determine the pain levels of cancer patients. | 2 months
  Pain levels for cancer patients
"Cancer Fatigue Scale" will be used to determine the fatigue levels of cancer patients. | 2 months
  Fatigue levels for cancer patients
"Rhodes nausea-vomiting and retching index" will be used to determine the nausea-vomiting levels of cancer patients. | 2 months
  Nausea-vomiting levels for cancer patients
"Spiritual Well-Being Scale" will be used to determine the spiritual well-being levels of cancer patients. | 2 months
  Spiritual well being levels for cancer patients

IPD SHARING:
Plan to Share IPD: No